CLINICAL TRIAL: NCT07097883
Title: The Impact of Previous Open Renal Surgery on Percutaneous Nephrolithotomy Complications
Brief Title: Impact of Previous Open Renal Surgery on Percutaneous Nephrolithotomy Complications
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Reyad, Assistant Professor of Urology, Faculty of Medicine, Sohag University, Sohag, Egypt, Sohag University
Other Study IDs: Soh-Med-25-6-1PD
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Open Renal Surgery; Percutaneous Nephrolithotomy; Complications
MeSH Terms: interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh cases: Patients with no prior renal surgery.
  Interventions: Procedure: Percutaneous Nephrolithotomy
- Recurrent cases: Patients with previous open renal surgery on the same side.
  Interventions: Procedure: Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous Nephrolithotomy — Patients underwent percutaneous nephrolithotomy (PCNL) for renal calculi >2 cm.

SUMMARY:
This study compared percutaneous nephrolithotomy (PCNL) complications in cases with or without previous renal surgery.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is a cornerstone in managing large renal calculi. However, in patients with a history of previous open renal surgery (POS), retroperitoneal scarring, altered anatomy, and vascular complications may influence PCNL outcomes.

The literature remains inconsistent regarding whether POS negatively impacts PCNL success or increases complications. Therefore, this study aims to clarify the comparative safety and efficacy of PCNL in patients with and without prior open renal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years).
* Both sexes.
* Undergoing percutaneous nephrolithotomy (PCNL) for renal calculi >2 cm.

Exclusion Criteria:

* Active urinary tract infection.
* Elevated serum creatinine >2.0 mg/dL.
* Pregnancy.
* Uncontrolled coagulopathy.
* Significant cardiopulmonary comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective hospital-based comparative study included 200 patients with recurrent renal stones in one arm and an equal number of patients in a control arm.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Hospital stay duration | Till the discharge from hospital (Up to two weeks)
  Lenght of hospital stay was recorded from the admission till the discharge from hospital.

SECONDARY OUTCOMES:
Serum creatinine level | Preoperatively
  Serum creatinine level was recorded.
Incidence of patients who need for auxiliary procedure | 24 hours postoperatively
  Incidence of patients who need for auxiliary procedure were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.